CLINICAL TRIAL: NCT04770857
Title: Evaluation of Post-Post-Endoscopic Retrograde Cholangiopancreaticography Pain (ERCP) as a Predictor for Post-ERCP Pancreatitis
Brief Title: Evaluation of Post-ERCP Pain as a Predictor for Post-ERCP Pancreatitis
Acronym: PEP-PREPARE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Nicola Frei (Other)
Responsible Party: Sponsor-Investigator, Nicola Frei, MD, Cantonal Hospital of St. Gallen
Organization: Cantonal Hospital of St. Gallen (Other)
Other Study IDs: CTU 19/036
Record Dates: First submitted 2021-02-22; First posted 2021-02-25 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Post-ERCP Acute Pancreatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Visual analogue scale — Post procedural pain assessment using the visual analogue scale (VAS) will be performed in patients undergoing ERCP

SUMMARY:
Pancreatitis is the most common complication after ERCP, although its frequency varies significantly depending on the study from < 2% up to 40%.

Based upon data from studies that have included unselected patients, post-ercp pancreatitis (PEP) is mild, moderate, and severe in 45%, 44%, and 11% of cases, respectively. Dysfunction of the sphincter Oddi, female gender, younger age, previous history of pancreatitis, prolonged procedure time and pancreatic guidewire passages are well-known independent risk factors for PEP.

This study will assess whether the development of PEP can be predicted by Visual analogue scale (VAS) level 1 hour after ERCP.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Scheduled for ERCP for any reason

Exclusion Criteria:

* Absence of consent
* Language barrier
* No endoscopic advance to the papilla vateri
* Active pancreatitis at the time of the procedure
* Mental disability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients scheduled for ERCP for any reason at the study center will be asked for participation.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Association between Pain 1 hour after ERCP | 1 hour

SECONDARY OUTCOMES:
Predictive value of VAS for PEP Predictive value of VAS for PEP | 1 hour
Association between VAS level and severity of PEP | 1 hour

CONTACTS AND LOCATIONS:
Locations (1):
- Kantonsspital Sankt Gallen, Sankt Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided